CLINICAL TRIAL: NCT04279275
Title: Degree of Knowledge About Anaesthesiology and Anaesthesiologists Among Patients in Tertiary Care Hospital of Kingdom of Saudi Arabia.
Brief Title: Knowledge About Anaesthesiology and Anaesthesiologists
Status: Completed | Type: Observational
Sponsor: Our Lady of Lourdes Hospital, Drogheda (Other Government)
Responsible Party: Principal Investigator, SHANKAR LAL, Primary Investigator, Our Lady of Lourdes Hospital, Drogheda
Other Study IDs: NGHA1
Record Dates: First submitted 2019-10-26; First posted 2020-02-21 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Knowledge; Anaesthesiology
Keywords: Field of Anaesthesiology; Knowledge; Survey
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Survey: Knowledge survey
  Interventions: Other: SURVEY

INTERVENTIONS:
Other: SURVEY — QUESTIONAIRRE

SUMMARY:
Object: To determine the Knowledge about anaesthesiologist's role and responsibilities along with the field of anaesthesiology among patients.

Study Design: A Cross-Sectional Survey. Place and Duration of Study: National Guard Health Affairs, from 1st December 2017 to 30th March 2018.

Methodology: After informed consent patients were asked to answer the questionnaire comprising of 12 open-ended questions regarding their knowledge about anaesthesiologist and anaesthesiology. Scoring as per correct and incorrect questions was done using version 19 (SPSS Inc., Chicago, IL).

DETAILED DESCRIPTION:
INTRODUCTION:

Anaesthesiology is still an emerging specialty in comparison to medicine and the field of surgery. Unawareness, infrequent exposure, and limited direct patient interaction have resulted in into least knowledge regarding the field of anaesthesiology among patients get admission to the hospital. The role, status of the anaesthesiologist and the awareness about the specialty of anaesthesiology has always been an active issue in the general population of most of the countries. Ongoing advancement in the field of anaesthesiology has facilitated complex surgical procedures, but it has never been acknowledged anywhere in media. Several studies done on the same subject is a reflection of efforts of professional bodies around the world towards improvement in the spread of awareness about the field of anaesthesiology and role of anaesthesiologist but these are still largely inaccurate.

A survey done even in developed countries outside the operating rooms depicted that the patients have limited awareness about the role of anaesthesiologists. A survey was done in India in 2018 showed that there was widespread ignorance about the anaesthesiology and role of anaesthesiologist in patients attending rural healthcare facilities. A 2009 survey in government busy setting of India showed that only 56% of patients knew that anaesthesiologist is a doctor. A survey done in the year 2004 revealed a high number of around 80% of patients visiting hospital recognized anaesthesiologist as a doctor but were unaware of their responsibilities in the hospital.

In the era of the rise in media and the Internet, an enhancement can be seen in awareness about anaesthesiology. Awareness about anaesthesiology and anaesthesiologists is an important better relationship between patient and doctor.

Methodology:

A cross-sectional study was conducted at the National Guard Health Affairs, Riyadh, Saudi Arabia from 1st December 2017 to 30th March 2018. The sample size was calculated using the WHO Sample Size Calculator. In a previous study, knowledge regarding anaesthesiologists and anaesthesiology was about 51.52% therefore 384 patients will be included in this study to estimate knowledge within 5 percent point (margin of error) of the true value (51.52%) with 95% confidence interval. Using Non-probability purposive sampling patients falling in inclusion criteria were included after taking ethical committee approval and patient's consent. Patients of either gender aged 18 to 60 years were included regardless of the specialty of surgery. We excluded those patients who refused to give consent and those were unable to give consent because of being language bearer, mentally not bill to understand questionnaires and doctors who were admitted as patients. Knowledge about anaesthesiologists and the field of anaesthesiology was measured by asking the questionnaire comprising 12 questions. Patients were interviewed by the preoperative anaesthetist and principal investigator on the ward. Each interview lasted for 10-20min and was based on a questionnaire in English and Arabic language. The questionnaire consisted of questions modified from previous studies and added questions. It had two parts; demographics i.e. age, gender, educational level, occupation, previous anaesthesia experience and type of surgery, the second part will consist of 12 questions about anaesthesiology and anaesthesiologist. Patients giving the correct responses to 8 out of 12 questions were considered to have knowledge. Data were analyzed using statistical packages for social science version 19 (SPSS Inc., Chicago, IL). Frequency and percentage were computed for gender, type of surgery, education level, previous surgery, Patient's knowledge about anaesthesiology and anaesthesiologist. Mean and the standard deviation was estimated for age. Stratification was done to control effect modifiers like gender, age, education level, previous surgery to observed the Patient's knowledge about anaesthesiology and anaesthesiologist through the chi-square test. p≤0.05 is considered as significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted in national guard health affairs.
* Age 18 and above.
* Both male and female

Exclusion Criteria:

* People refusing to give consent.
* Pediatric patients (patients up to age of 16 years).
* Language barrier.
* Patient unable to understand the questions due to disability.
* Patients who are doctors.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult Patients
Sampling Method: Non-Probability Sample
Enrollment: 385 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
Number of participants having knowledge about field of anaesthesiology and role of anaesthetist assessed with questionnaire. | 1 year
  Patients Giving Correct answers of 8 Questions Out Of 12 on questionnaire will be Labelled having sufficient Knowledge. If the Total Number of Correct answers is less than 8 out of 12, it will be considered Insufficient Knowledge about Anaesthesiology and Role of Anaesthetists.

CONTACTS AND LOCATIONS:
Overall Officials: SHANKAR LAL, MBBS/FCPS, Principal Investigator — Our Lady of Lourdes Hospital
Locations (1):
- Our Lady of Lourdes Hospital, Drogheda, Louth, Ireland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Singh T, Sharma S, Banerjee B, Garg S. Knowledge regarding anesthesiologist and anesthesiology among patients and attendants attending a rural hospital of New Delhi. J Educ Health Promot. 2018 Jan 10;7:12. doi: 10.4103/jehp.jehp_52_17. eCollection 2018. PMID 29417072
- [Result] Jindal P, Khurana G, Bharadwaj A, Mallik S, Oberoi D. Current understanding of the literate versus illiterate patient's knowledge about anesthesiologists: A comparative study. Anesth Essays Res. 2013 Jan-Apr;7(1):58-64. doi: 10.4103/0259-1162.113994. PMID 25885722
- [Result] Lee JJ, Lee NH, Park CM, Hong SJ, Kong MH, Lee KH, Yon JH, Song SO. Public awareness about the specialty of anesthesiology and the role of anesthesiologists: a national survey. Korean J Anesthesiol. 2014 Jan;66(1):12-7. doi: 10.4097/kjae.2014.66.1.12. Epub 2014 Jan 28. PMID 24567807